CLINICAL TRIAL: NCT06673225
Title: Evaluation of the Implementation of the INSPIRE Respiratory Health Program: Integration of Early Diagnosis and Emergency Response for Respiratory Diseases in the City of Botucatu, São Paulo, Brazil
Brief Title: INSPIRE Respiratory Health Program in Botucatu, São Paulo, Brazil
Status: Recruiting | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Other Study IDs: Inspire2024
Record Dates: First submitted 2024-07-15; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Community Health Services; Respiratory Disease; Tobacco Smoking
Keywords: Primary care; Health promotion; Pulmonary function tests; Nicotine addiction; Smoking cessation
MeSH Terms: conditions — Respiration Disorders; Tobacco Smoking; Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single group: History of smoking and/or passive exposure and/or respiratory symptoms.
  Interventions: Other: Analysis of results

INTERVENTIONS:
Other: Analysis of results — Analysis of previous imaging and/or laboratory tests, vital signs, body composition, pulmonary function, peripheral muscle strength, calf circumference, nutritional risk, quality of life, frailty level, and anxiety and depression. Screening for respiratory diseases, including chronic obstructive pulmonary disease (COPD), lung cancer, tuberculosis, and other lung lesions, is based on spirometry and thoracic radiological images after the health professional's examination. After the multiprofessional procedures, patients will be evaluated by a physician to start specific treatment and/or perform complementary exams if necessary. Every year, they will be re-evaluated to record acute exacerbations of chronic respiratory diseases and assess disease progression through spirometry and thoracic radiological images.

SUMMARY:
The goal of this observational study is to evaluate the implementation of the INSPIRE program and to plan actions for the preparation, coordination, monitoring, diagnosis, and treatment of respiratory diseases in the municipality of Botucatu. Methods: Individuals with respiratory symptoms from the municipality of Botucatu, aged 18 or older, will be invited to participate in the study, and socioeconomic data, as well as information on sex, gender, race, nutritional risk, frailty, tobacco exposure, and its derivatives, will be collected. For those with exposure, screening and treatment for respiratory diseases will be offered through assessment of pulmonary function, body composition, respiratory and peripheral muscle strength. Additionally, individuals over 40 years old with tobacco exposure equal to or greater than 30 pack-years will be offered low-dose chest CT screening for lung cancer. Expected results: To identify and assess vulnerable groups that face difficulties in accessing respiratory healthcare, as well as implement specific strategies for the treatment of respiratory diseases and tobacco control for these groups. To ensure equitable access to respiratory health for the entire population at risk due to smoking. Moreover, through proactive and reactive risk reduction actions implemented by the program, to intervene in distinct groups and other regions.

DETAILED DESCRIPTION:
The project focuses on evaluating the management in the implementation of the INSPIRE respiratory health program, being applied in the health network of the municipality of Botucatu with the active co-participation of municipal managers and the local population, aiming to achieve all the proposed results. This thorough evaluation will be conducted through a longitudinal cohort study, with patient follow-up over five years. All evaluated subjects will be contacted annually to contribute to effective management and positive outcomes in respiratory health. The primary care networks (basic health and family health networks), secondary care, including urgent care and emergency units, and tertiary health care in Botucatu (tertiary hospital in the municipality of Botucatu) will participate.

The local media and primary health care unit will be informed of the monthly dates on which individuals with a history of smoking and/or passive exposure and/or respiratory symptoms can be referred for a multiprofessional evaluation. This referral can be made during a consultation or by spontaneous demand at the primary health care unit, which in turn will refer for specialized evaluation.

Statistical analyses will be divided into three main packages: disease incidence, clinical evaluation, and AI algorithms. Positive cases occurring during the evaluation period will be considered for disease incidence. For incidence calculation, the time to diagnosis for each participant will be considered in a measure expressed in person-years. Poisson regression models will be applied to estimate the relative risk for incidence among all possible groups to compare sociodemographic and other characteristics. Adjustments for possible confounding factors may be necessary and will be decided later. The second package includes the comparison between clinical characteristics and body composition. Positively and negatively screened individuals will be compared using appropriate statistical tests. Continuous variables will be tested for symmetry, and appropriate tests will be conducted (t-test or Wilcoxon; ANOVA or Mann-Whitney; parametric or non-parametric regression models). Fisher's exact tests and Chi-square (heterogeneity or trends) will be used for categorical variables.

Each participant will have their coding, preventing the identification of patients. Medical data will be kept confidential and securely stored. To ensure data quality, all researchers will be trained before the start of the study, contact with the coordinator will be allowed to clarify study protocol-related doubts, coded electronic databases will be used, which will be monitored by an external team to the study and will draw patient codes that will be monitored and their data certified. Discrepant data will automatically question the veracity of the data to reduce data inconsistency. Data will be continuously monitored to identify and correct inconsistencies. The data capture program will be REDCap, in which the developer will be solely responsible for database modifications after approval by the scientific committee.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years old;
* Respiratory symptoms
* History of active or passive smoking
* Signing of informed consent form

Exclusion Criteria:

* Difficulty understanding the issues addressed
* Inability to contact by phone
* Non-signing or withdrawal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with a history of smoking and/or passive exposure and/or respiratory symptoms residing in the city of Botucatu, state of São Paulo, Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2029-04-15 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of changes in respiratory disease incidence following the implementation of the INSPIRE Program in Botucatu | One year
  This primary outcome assesses the program's effectiveness in public health by directly measuring changes in the incidence of respiratory diseases within the target population

SECONDARY OUTCOMES:
Program implementation costs | One year
  This measure estimates the total costs associated with implementing the program. It includes all expenditures related to program activities and administration.

CONTACTS AND LOCATIONS:
Overall Officials: Suzana E Tanni, MD-PhD, Principal Investigator — São Paulo State University (UNESP), Medical School, Botucatu
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Botucatu, Botucatu, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No